CLINICAL TRIAL: NCT00286533
Title: Retrospective Evaluation of Implants Placed in the Regular Dentist's Practice. A Study to Evaluate Implant Success, Prosthetic Complications, Opinion of the Patient, and Quality of Care
Brief Title: Evaluation of Implants Placed in the Regular Dentist's Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/414
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Dental Implant
Keywords: Implant
MeSH Terms: interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placed implants (Experimental)
  Interventions: Procedure: Clinical examination (implant stability, gingiva condition, etc.); Procedure: Questionnaires

INTERVENTIONS:
Procedure: Clinical examination (implant stability, gingiva condition, etc.) — Clinical examination (implant stability, gingiva condition, etc.) to follow
Procedure: Questionnaires — Questionnaires are used.

SUMMARY:
This study is an evaluation of the implants placed in a regular dentist's practice regarding:

* gingiva condition
* stability of implant
* prothetic quality
* questionnaires for the patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with implants placed in a regular dentist's practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
gingiva condition | t0

OTHER OUTCOMES:
stability of implant | t0
prothetic quality | t0
questionnaires for the patients | t0

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be